CLINICAL TRIAL: NCT00101959
Title: An Implementation Study of Treatment Optimization Recommendations Comparing Subjects Continuing Treatment With IFN-ß-1a 30 Mcg qw IM (Avonex®) or Glatiramer Acetate 20 mg qd SC (Copaxone®) to Those Randomized to IFN-ß-1a 44 Mcg Tiw SC (Rebif®), in a Multicenter Study of Subjects With Relapsing Remitting Multiple Sclerosis Currently on Disease-Modifying Therapy
Brief Title: Implementation Study of Treatment Optimization Recommendations on Relapsing-Remitting Multiple Sclerosis (RR MS) Subjects
Status: Withdrawn | Phase: Phase 4 | Type: Interventional
Sponsor: EMD Serono (Industry)
Responsible Party: Sponsor
Purpose: Treatment
Other Study IDs: 25277
Record Dates: First submitted 2005-01-18; First posted 2005-01-19 (Estimated); Last update posted 2013-08-06 (Estimated); Status verified 2013-08

CONDITIONS: Relapsing-Remitting Multiple Sclerosis
MeSH Terms: conditions — Multiple Sclerosis, Relapsing-Remitting | interventions — Interferon beta-1a

INTERVENTIONS:
Drug: Rebif

SUMMARY:
Brief Summary: 800 RRMS Subjects currently treated with Avonex or Copaxone will be randomized to either continue on their current therapy or receive Rebif therapy. The subjects will be followed for 2 years. The primary objective is to compare the time to worsening to a medium level of concern as defined by the Canadian Multiple Sclerosis Working Group (CMSWG) treatment optimization recommendations.

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent (and HIPAA authorization for USA subjects) before any study-related procedure, not part of the subject's normal medical care, with the understanding that the subject could withdraw consent at any time without prejudice to future medical care
* Age between 18 and 60 years (inclusive)
* Male and female subjects with clinically definite or laboratory-supported definite relapsing-remitting multiple sclerosis based on Poser or McDonald criteria
* Results of an MRI scan acquired within 2 years of screening, consistent with MS.
* Duration of MS ≤ 7 years from onset of symptoms
* Receiving consistent therapy with Avonex®, or Copaxone® for ≥ 2 years (Subjects that have converted from one therapy to another or who have used other disease-modifying therapies (DMTs) within two years of Screening will be excluded).
* Expanded Disability Status Score (EDSS) of 0 to ≤ 5.5, inclusive
* Exhibiting low or medium level of concern based on number and severity of relapses within 12 months prior to screening (subjects who have reached a high level of concern at any time within the past 12 months will be excluded); *Low Level of Concern: a) 1 mild relapse (Mild severity - corticosteroids not required, minimal effect on Activities of Daily Living (ADL), only 1 Kurtzke Functional Systems (KFS) functional domain affected, no or mild motor/cerebellar involvement, no need for treatment or hospitalization and prompt recovery); *Medium Level of Concern: a) 2 mild relapses or 1 moderate relapse (Moderate severity - corticosteroids may be required, at most moderate effect on ADL, >1 KFS functional domain may be affected, moderate motor/cerebellar involvement, may require treatment but not hospitalization and incomplete recovery at 3 months but complete recovery by 6 months)
* Clinical stability or improving neurological state during the eight weeks before Study Day 1
* Willingness and ability to comply with the protocol for the duration of the study
* If female, she must either:

  1. be post-menopausal or surgically sterilized; or
  2. use a hormonal contraceptive, intrauterine device, diaphragm with spermicide, or condom with spermicide, for the duration of the study; and
  3. be neither pregnant nor breast-feeding.
  4. confirmation that the subject is not pregnant must be established by a negative serum hCG pregnancy test within 30 days of Study Day 1 and a negative urine pregnancy test on Study Day 1. A pregnancy test is required for all females that are of childbearing potential.
* The small minority of subjects for whom Rebif therapy is not reimbursed by their insurance carrier may be considered for the study if otherwise eligible, but will require prior approval from the sponsor for coverage of the cost of their Rebif therapy

Exclusion Criteria:

* Pregnant or lactating women, or women of childbearing potential not using an acceptable method of contraception
* Progressive forms of MS (Primary progressive, Secondary progressive)
* Exhibiting a high level of concern based on number and severity of relapses at any time in the 12 months prior to screening; *High Level of Concern a) 3 mild, 2 moderate or 1 severe relapse (Severe Severity- Corticosteroids and hospitalization required, severe effect on ADL, >1 KFS functional domain may be affected, severe motor/cerebellar involvement, impact on ADL and incomplete recovery at 6 months)
* Subjects who have been on DMTs other than Avonex® or Copaxone® in the two years prior to screening.
* Subjects with history of intolerance to Interferon Beta
* History of hypersensitivity to natural or recombinant interferon beta, human serum albumin, or any other component of the Rebif® formulation including mannitol
* History of hypersensitivity to natural or recombinant interferon beta, human serum albumin, or any other component of the Rebif® formulation including mannitol
* Participation in any other studies involving investigational or marketed products, concomitantly or within 3 months prior to Study Day 1
* Treatment with oral or systemic corticosteroids or ACTH within 4 weeks of Study Day 1 or ongoing chronic treatment with systemic corticosteroids.
* Treatment with immunomodulatory or immunosuppressive therapy (including but not limited to cyclophosphamide, cyclosporine, methotrexate, azathioprine, linomide, mitoxantrone, Campath) within the 12 months prior to Study Day 1
* Prior cytokine or anti-cytokine therapy within 3 months prior to Study Day 1
* Prior use of cladribine or have received total lymphoid irradiation
* Prior use of Antegren® (natalizumab)
* Have taken intravenous immunoglobulin or any other investigational drug or taken part in any experimental procedure in the 3 months prior to Study Day 1
* Psychiatric disorder that is unstable or would preclude safe participation in the study
* Cognitive impairment which impairs ability to understand or comply with the protocol procedures
* Any laboratory value reaching Grade 2 toxicity or greater within 30 days of Study Day 1 based on Common Terminology Criteria for Adverse Events (CTACE) criteria
* Specific systemic diseases, (including insulin-dependent diabetes, Lyme disease, clinically significant cardiac disease, HIV, HTLV-1, and Hepatitis B or C), or other uncontrolled major medical conditions (depression, seizure disorder) that would interfere with the participant's safety, compliance or evaluation
* Unable and/or unlikely to follow the protocol for any reason
* Alcohol and/or any other drug abuse
* Likelihood of requiring treatment during the study period with drugs not permitted by the study protocol
* Abnormal baseline clinical findings considered by the investigator to be indicative of conditions that might affect study results

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 0 (Actual)
Dates: Start 2004-11

REFERENCES:
- See also: Full FDA approved prescribing information can be found here — http://www.mslifelines.com